CLINICAL TRIAL: NCT06750913
Title: PCNL Without Reverse Catheterization in the Split-leg Prone Position: A Randomized Controlled Trial.
Brief Title: PCNL Without Reverse Catheterization in the Split-leg Prone Position.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Director, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Guohua Zeng
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Urinary Stones
MeSH Terms: conditions — Urinary Calculi | interventions — Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In the study group, the patient is directly placed in the split-leg prone position. A 10-cm soft pillow is used to elevate the upper abdomen, making the lower edge of the pubic symphysis exceed the lower edge of the operating table by 5 cm. The patient's legs are spread in a V-shaped manner. The thigh on the healthy side is abducted as much as possible, while the thigh on the affected side is slightly abducted, so that the angle between the two legs is approximately 80°. The lumbar back and perineum are disinfected and covered with sterile drapes, and an indwelling urinary catheter is inserted for open drainage. The target renal calyx is punctured percutaneously under the guidance of ultrasound, and an 18 - 24 Fr tract is established under the guidance of a guidewire. A peel-away working sheath is then left in place, completing the establishment of the tract.
  Interventions: Procedure: Comparison between PCNL without Catheterization in the Split-leg Prone Position and Traditional PCNL
- Control group (No Intervention): In the control group, the patient is first placed in the lithotomy position. A 5 Fr ureteral catheter is retrogradely inserted into the ureter on the affected side via a cystoscope, along with a 16 Fr Foley catheter. Then, the patient is turned to the prone position, and a 10-cm soft pillow is used to elevate the upper abdomen. The surgical area is disinfected and draped again. Sterile normal saline is injected through the ureteral catheter to create artificial hydronephrosis. The target renal calyx is punctured percutaneously under the guidance of ultrasound, and retrograde contrast is performed when necessary, combined with X-ray-guided percutaneous puncture. Subsequently, an 18 - 24 Fr tract is established under the guidance of a guidewire, and a peel-away working sheath is left in place, thus completing the establishment of the tract.

INTERVENTIONS:
Procedure: Comparison between PCNL without Catheterization in the Split-leg Prone Position and Traditional PCNL — Before the start of PCNL, one group of patients was placed in the lithotomy position and then converted to the prone position, and one group of patients directly separated from the leg prone position without an external brace
  Arms: Experimental group

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is currently the first-line treatment for upper urinary tract stones larger than 2 cm. It is minimally invasive and enables rapid recovery, thus winning the approval of patients . In the traditional PCNL procedure, a ureteral catheter is first retrogradely inserted into the ureter on the affected side with the patient in the lithotomy position, and then the patient is changed to the prone position for percutaneous renal puncture and stone extraction . The inserted catheter can be used for retrograde injection of water or contrast agents, which facilitates percutaneous renal puncture and also prevents stone fragments from entering the ureter during the lithotripsy process . However, under the lithotomy position, disinfection, draping, and intubation are carried out first, and then the patient is turned to the prone position for another round of disinfection and draping, which is cumbersome and requires a long surgical preparation time.

In recent years, with the enrichment of urologists' experience in percutaneous renal puncture and the improvement of the quality of ultrasound images, the application of percutaneous renal puncture and fistulization guided by ultrasound has become more and more widespread . Experienced urologists can even puncture the target renal calyx without the need for retrograde intubation and injection of water to form an "artificial hydronephrosis". Combined with intraoperative contrast verification through the puncture needle, accurate puncture can be ensured. This saves the surgical time required for the traditional PCNL, which involves retrograde intubation in the lithotomy position followed by a change to the prone position, and also avoids the risk of infection that may be increased due to elevated renal pelvic pressure during retrograde injection. However, failure to place a retrograde catheter during PCNL may increase the difficulty of puncture and the risk of stone fragments entering the ureter during the lithotripsy process. We adopt the split-leg prone position, and when necessary, retrograde ureteroscopic operations can be performed. In this way, various needs for anterograde and retrograde operations can be met in a single position .

Direct percutaneous renal puncture and stone extraction under the guidance of ultrasound combined with X-ray without retrograde intubation in the split-leg prone position has both advantages and disadvantages, posing a challenge to surgeons. To verify the safety and feasibility of this technique, we have launched this clinical randomized controlled trial for verification.

DETAILED DESCRIPTION:
### 1. Research Background Percutaneous nephrolithotomy (PCNL) is currently the first-line treatment for upper urinary tract stones larger than 2 cm. It is minimally invasive and enables rapid recovery, so it has gained patients' approval. When performing PCNL, most urologists first place a ureteral catheter retrogradely into the ureter on the affected side with the patient in the lithotomy position, and then change the patient to the prone position for percutaneous renal puncture and stone extraction. The retrogradely inserted catheter can be used for injecting water or contrast agents in reverse, which facilitates percutaneous renal puncture and also prevents stone fragments from entering the ureter during the lithotripsy process. However, when performing PCNL in the standard prone position, it may sometimes be difficult to place an anterograde internal stent or treat ureteral stones, requiring the patient to be changed back to the lithotomy position again. This entails another round of disinfection and draping, thus increasing the workload of the medical team and prolonging the operation time.

In recent years, with urologists gaining more experience in percutaneous renal puncture and the improvement of the quality of ultrasound images, the application of ultrasound-guided percutaneous renal puncture and fistulization has become increasingly popular, being no less effective than X-ray. Ultrasound-guided percutaneous renal puncture and fistulization does not rely on retrograde pyelography. Even experienced urologists do not need to perform retrograde intubation and water injection to form an "artificial hydronephrosis", which saves the operation time required for the traditional procedure of retrograde intubation in the lithotomy position followed by changing to the prone position, and also avoids the risk of infection caused by the possible increase in renal pelvic pressure during retrograde water injection. However, not placing a retrograde catheter may lead to difficulties in puncturing a non-hydronephrotic kidney. During the PCNL lithotripsy process, if stone fragments enter the ureter and are difficult to manage anterogradely, retrograde ureteroscopic treatment is required again, which is difficult to perform in the traditional simple prone position and requires changing back to the lithotomy position. In fact, retrograde ureteroscopic operations can be carried out in the split-leg prone position, which can meet various requirements for anterograde and retrograde operations during PCNL in a single position. This is the particular advantage of PCNL in the split-leg prone position.

Direct percutaneous renal puncture and stone extraction under ultrasound guidance without retrograde intubation in the split-leg prone position can save the operation time of the traditional procedure of intubation in the lithotomy position followed by changing to the prone position. However, there is a risk of stone fragments entering the ureter during lithotripsy. This can be addressed by retrograde ureteroscopy in the split-leg prone position. In addition, higher technical requirements are imposed on ultrasound-guided percutaneous renal puncture. Whether this technique is feasible still needs to be clinically verified.

* 2. Research Objectives To conduct a single-center, prospective, randomized, controlled study to explore the safety, feasibility, and potential advantages of percutaneous nephrolithotomy without retrograde intubation in the split-leg prone position.

  * **Primary outcome measures**: The time to establish the first tract, operation time.
  * **Secondary outcome measures**: Stone-free rate, surgical complications.
* 3. Research Design

  * **3.1 Research nature**: A single-center, randomized, controlled trial with a 1:1 two-group parallel design, which is randomized and open-label.
  * **3.2 Sample size**: According to the literature and preliminary experiments, the operation times for percutaneous nephrolithotomy without a ureteral catheter in the split-leg prone position and in the traditional position for treating 2 - 5 cm renal stones are (71.95 ± 21.11) minutes and (95.01 ± 25.06) minutes respectively. Assuming that the operation time of PCNL without a ureteral catheter in the split-leg prone position is shorter than that of traditional PCNL, with a type-1 error (α) of 0.05, a power (1 - β) of 0.8, a 1:1 ratio of the two groups, and a superiority test boundary value of - 10, the required sample size for Fisher's exact test for comparing the two groups is calculated according to the Walters approximation algorithm. Forty patients are required for each group. Considering issues such as dropouts, the sample size of each group is expanded to 45, with a total of 90 patients enrolled.
  * **3.3 Random grouping and control methods**: This study adopts a balanced randomization method to generate a random number table and randomly assign patients to groups. The trial uses a mutual control method. Group 1 is the split-leg prone position without a ureteral catheter group, and group 2 is the traditional group. Specific interventions: 1. The surgical position of group 1 is the split-leg prone position, while that of group 2 is first the lithotomy position and then the prone position; 2. Group 1 does not place a ureteral catheter retrogradely, while group 2 does.
* 4. Research Subjects A total of 90 patients with 2 - 7 cm upper urinary tract stones.

  * **Inclusion criteria**: 1. Agree to participate in this RCT; 2. Aged 18 - 70 years; 3. Upper urinary tract stones 2 - 7 cm.
  * **Exclusion criteria**: 1. Those who have already undergone nephrostomy or second-stage surgery; 2. Patients with abnormal anatomical structures, such as ectopic kidney, horseshoe kidney, duplex kidney, transplanted kidney, etc.; 3. Pregnant women; 4. Incomplete data or lost to follow-up.
  * **Withdrawal criteria for subjects**: If purulent fluid is found during intraoperative puncture, a nephrostomy tube will be placed and the operation will be terminated, and the patient will be excluded from the group; patients may also withdraw voluntarily.
* 5. Research Process

  * **5.1 Preoperative examinations**:
  * **(1) Laboratory tests**: Complete blood count, routine urine test, midstream urine culture, liver and kidney function tests, electrolyte tests, coagulation function tests, and blood-borne disease screening.
  * **(2) Imaging examinations**: Unenhanced CT scan of the urinary system, KUB, chest X-ray, electrocardiogram, and echocardiogram if necessary.
  * **5.2 Preoperative preparation**:
  * For patients with a positive preoperative urine culture, sensitive antibiotics should be selected according to the drug sensitivity test to control the infection for 5 - 7 days. For patients with a negative preoperative urine culture, a single dose of broad-spectrum antibiotics is given prophylactically.
  * One day before the operation, eligible patients are enrolled according to the generated random number table and number, and the informed consent form is signed. Patients corresponding to "0" in the random number table are arranged into the study group (group 1) to undergo PCNL without a ureteral catheter in the split-leg prone position; those corresponding to "1" are arranged into the control group (group 2) to undergo PCNL in the traditional position.
  * **5.3 Surgical methods**:
  * All patients receive general anesthesia with endotracheal intubation.
  * In the study group, the patient is directly placed in the split-leg prone position. A 10-cm soft pillow is used to elevate the upper abdomen, with the lower edge of the pubic symphysis exceeding the lower edge of the operating table by 5 cm. The patient's legs are spread in a "V" shape. The thigh on the healthy side is abducted as much as possible, while the thigh on the affected side is slightly abducted, making the angle between the two legs approximately 80°. The lumbar back and perineum are disinfected and draped, and a urinary catheter is inserted for open drainage. Ultrasound is used to guide the percutaneous puncture of the target renal calyx, and an 18 - 24 Fr tract is established under the guidance of a guidewire, with a peel-away working sheath placed to complete the tract establishment.
  * In the preoperative group, the patient is placed in the lithotomy position. A 5 Fr ureteral catheter is retrogradely inserted into the ureter on the affected side through a cystoscope, along with a 16 Fr Foley catheter. Then the patient is turned to the prone position, with a 10-cm soft pillow elevating the upper abdomen, and the surgical area is disinfected and draped again. Sterile normal saline is injected through the ureteral catheter to create artificial hydronephrosis. Ultrasound is used to guide the percutaneous puncture of the target renal calyx, and retrograde contrast is performed if necessary, combined with X-ray-guided percutaneous puncture. Subsequently, an 18 - 24 Fr tract is established under the guidance of a guidewire, with a peel-away working sheath placed to complete the tract establishment.
  * After the tract is established, a nephroscope is inserted through the working sheath of the tract, and pneumatic ballistic or holmium laser lithotripsy is performed under the irrigation of the perfusion pump, with a negative pressure suction sheath used to clean the stone fragments. After lithotripsy, bedside X-ray fluoroscopy is used to check the stone clearance status, and further treatment of residual stones is carried out if necessary. For migrated residual ureteral stones that are difficult to manage anterogradely, retrograde ureteroscopy is performed in the split-leg prone position in the study group, while in the control group, the patient is turned to the lithotomy position, disinfected and draped again, and then retrograde ureteroscopy is carried out. Whether to place an internal stent and a nephrostomy tube is determined according to the surgical situation. If there are no active stone residues, no ureteral obstruction, no significant bleeding in the tract, and no perforation or bleeding in the collecting system, a tubeless approach can be adopted. The operation is completed. All operations are performed by the same urologist.

ELIGIBILITY:
Inclusion Criteria:

* Consent to enter the RCT;
* Age 18-70 years old;
* Upper urinary tract stones 2-7cm;

Exclusion Criteria:

* Those who have undergone nephrostomy and second-stage surgery;
* Patients with abnormal anatomical structures, such as ectopic kidneys, horseshoe kidneys, duplicate kidneys, transplanted kidneys, etc.;
* Pregnant women;
* Incomplete or lost to follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
The first channel establishment time | 1 week
Duration of surgery | Intraoperative

SECONDARY OUTCOMES:
Stone clearance rate | 1 week
Complications of surgery | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China